CLINICAL TRIAL: NCT04722172
Title: A Phase 2 Time Limited Approach Based on Depth of Response to Front-Line Acalabrutinib in Combination With Obinutuzumab for CLL/SLL Patients Who Achieve Complete Remission or Partial Remission With Undetectable Minimal Residual Disease
Brief Title: A Study on Limiting Treatment Time With Acalabrutinib Combined With Obinutuzumab in People With CLL or SLL
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: AstraZeneca (Industry); Genentech, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-503
Record Dates: First submitted 2021-01-20; First posted 2021-01-25 (Actual); Last update posted 2025-08-27 (Actual); Status verified 2025-08

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: Acalabrutinib; Obinutuzumab; 20-503
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — acalabrutinib; obinutuzumab

STUDY DESIGN:
Intervention Model Description: This is a phase II, multicenter clinical trial.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Acalabrutinib Combined With Obinutuzumab (Experimental): Patients will receive acalabrutinib for a minimum of 13 cycles and maximum 26 cycles and Obinutuzumab will be administered during Cycles 2-7. This will be followed by treatment-free observation through the 65th cycle. Patients who progress during the observation period, per iwCLL criteria, will receive 13 cycles of acalabrutinib in combination with obinutuzumab in the retreatment phase of this study.
  Interventions: Drug: Acalabrutinib; Drug: Obinutuzumab

INTERVENTIONS:
Drug: Acalabrutinib — Acalabrutinib for a minimum of 13 cycles and maximum 26 cycles.
Drug: Obinutuzumab — Obinutuzumab will be administered during Cycles 2-7.

SUMMARY:
This study will test the safety of limiting treatment time with acalabrutinib and obinutuzumab in people who have chronic lymphocytic leukemia (CLL) or small lymphocytic lymphoma (SLL). The researchers want to find out whether stopping the study drugs when the cancer responds to the treatment, followed by a period of observation in which no treatment is given, is better than, the same as, or worse than the usual approach. A usual treatment for CLL and SLL is to give the study drugs continuously until the cancer progresses, even if the disease is in remission. But when people receive these drugs for long periods of time, they can have serious side effects and their cancer can become resistant to treatment.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent form (ICF). Legally Authorized Representatives are permitted.
* Ability and willingness to comply with requirements of the study protocol
* ≥ 18 years-old
* Have documented previously untreated CLL or SLL per WHO criteria and require treatment per iwCLL guidelines
* ECOG performance status of 0, 1, or 2, with no deterioration over the previous 2 weeks prior to baseline or day of first dosing
* Participants must have adequate organ and marrow function as defined below:

  * Total bilirubin ≤ 1.5 times upper limit of normal (ULN), unless there is a disease involvement of the liver, hemolysis, or a known history of Gilbert's disease.
  * Hemoglobin ≥ 8 g/dL without transfusion support, unless anemia is due to marrow involvement of CLL.
  * Absolute neutrophil count (ANC) ≥ 1.0 x 10^9/L.
  * AST and ALT ≤ 2.5 times the ULN.
  * Creatinine clearance (CrCl) > 30 mL/min as calculated using modified Cockcroft- Gault or MDRD Formula
  * PT/INR ≤ 2 times the ULN and aPTT ≤ 2 times the ULN unless the elevation in PT/INR or aPTT is solely attributable to direct oral anticoagulant.
* Platelet count without transfusion support must be ≥ 50,000 cells/mm3 or ≥ 30,000 cells/mm^3 in subjects with documented bone marrow involvement, as determined locally.
* For women of childbearing potential: Agreement to remain abstinent (refrain from heterosexual intercourse) or use a highly effective contraceptive method (failure rate of < 1%) per year during the treatment period and for at least 18 months after the last dose of study medication. Women of childbearing potential must have a negative serum pregnancy test result within 3 days prior to initiation of study drug

  * Women must refrain from donating eggs during this same period
  * A woman is considered of childbearing potential if she is postmenarcheal, has not reached a postmenopausal state (≥ 12 continuous months of amenorrhea with no identified cause other than menopause), and has not undergone surgical sterilization (removal of ovaries and/or uterus)
  * Examples of contraceptive methods with a failure rate of < 1 % per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices
* Examples of contraceptive methods with a failure rate of < 1 % per year include bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices

  * With female partners of childbearing potential, men must remain abstinent or use a condom plus an additional contraceptive method that together result in a failure rate of < 1% per year during the treatment period and for at least 6 months after- the last dose of obinutuzumab; men must refrain from donating sperm during this same period
  * With pregnant female partners, men must remain abstinent or use a condom during the treatment period and for at least 6 months after the last dose of obinutuzumab to avoid exposing the embryo
  * The reliability of sexual abstinence should be evaluated in relation to the duration of the clinical trial and the preferred and usual lifestyle of the patient; periodic abstinence (e.g., calendar, ovulation, symptothermal, or post-ovulation methods) and withdrawal are not acceptable methods of contraception

Exclusion Criteria:

* Prior CLL-directed therapy

  °Excluding corticosteroid therapy started for non-CLL related reasons or brief courses for disease related symptom management
* Received any investigational drug within 30 days or 5 half-lives (whichever is shorter) before first dose of study drug
* History of prior malignancy that could affect compliance with the protocol or interpretation of results, except for the following:

  * Curatively treated basal cell carcinoma or squamous cell carcinoma of the skin or carcinoma in situ of the cervix or carcinoma in situ of the prostate at any time prior to study.
  * Other cancers not specified above that have been curatively treated by surgery and/or radiation therapy from which subject is disease-free for ≥3 years without further treatment.
* Transformation of CLL to aggressive lymphoma (Richter's transformation to NHL or Hodgkin's lymphoma, or pro-lymphocytic leukemia)
* CLL with deletion of chromosome 17p and/or TP53 mutation. Patients must have FISH or array CGH analysis and NGS for TP53 mutations locally as per SOC within 60 days of C1D1 (peripheral blood, bone marrow or lymph node with disease involvement are acceptable sources) as SOC.
* History of or ongoing confirmed central nervous system (CNS) lymphoma.
* Known hypersensitivity to any active ingredient in the study drugs.
* Active bleeding, or presence of known bleeding disorder (e.g. von Willebrand's disease) or hemophilia.
* Any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study such as:

  * Clinically significant cardiac disease that includes symptomatic arrhythmia (subjects with controlled, asymptomatic atrial fibrillation or other atrial arrhythmias during screening are allowed to enroll on study)
  * Intracranial hemorrhage, stroke within 6 months of study enrollment
  * Symptomatic, or history of documented congestive heart failure (NY Heart Symptomatic, or history of documented congestive heart failure (NY Heart Association functional classification III-IV
  * Myocardial infarction within 6 months of enrollment
  * Concomitant use of medication known to cause QT prolongation or torsade's de pointes should be used with caution and at investigator's discretion
  * Angina not well-controlled by medication
  * Poorly controlled or clinically significant atherosclerotic vascular disease including cerebrovascular accident (CVA), transient ischemic attack (TIA), angioplasty, cardiac/vascular stenting within 6 months of study enrollment
* Known active bacterial, viral, fungal, mycobacterial, parasitic, or other infection (excluding fungal infections of nail beds) at study enrollment, or any major episode of infection requiring treatment with IV antibiotics or hospitalization (relating to the completion of the course of antibiotics) within 2 weeks prior to cycle 1 day 1 including subjects with positive cytomegalovirus [CMV] DNA polymerase chain reaction [PCR].
* Requires the use of warfarin or equivalent Vitamin K antagonist
* Requires or received the following agents within 7 days prior to the first dose of acalabrutinib-obinutuzumab combination therapy:

  * Patients who are positive for HCV antibody must be negative for HCV by polymerase chain reaction (PCR) to be eligible for study participation
  * Patients with occult or prior HBV infection (defined as positive total hepatitis B core antibody [HBcAb] and negative HBsAg) may be included if HBV DNA is undetectable by PCR. These patients must be willing to undergo sequential DNA testing as per institutional standards (every 1-3 months) and antiviral prophylaxis as per institutional standards.
* Uncontrolled AIHA (autoimmune hemolytic anemia) or ITP (idiopathic thrombocytopenic purpura).
* Presence of a gastrointestinal ulcer diagnosed by endoscopy within 3 months before screening, this is subject to investigator's discretion
* Known infection with HIV (testing not required as part of screening)
* Receipt of live-virus vaccines within 28 days prior to the initiation of study treatment
* Pregnant or lactating, or intending to become pregnant during the study
* Major surgical procedures within 28 days of first dose of study drug. Note: if a subject had major surgery, they must have recovered adequately from any toxicity and/or complications from the intervention before the first dose of study drug.
* Malabsorption syndrome or other condition that precludes enteral route of administration; this is subject to investigator discretion
* Has difficulty with or is unable to swallow oral medication
* Concurrent participation in the treatment phase of an interventional clinical trial
* Unwilling or unable to participate in all required study evaluations and procedures. Unable to provide a signed and dated informed consent form (ICF) and authorization to use protected health information (in accordance with national and local patient privacy regulations).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2021-05-21 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
progression-free survival (PFS) | 36 months
  Progression free survival (PFS) will be measured from the time the patient initiates treatment, until documented progression of disease, relapse, or death due to any cause, whichever comes first.

SECONDARY OUTCOMES:
Adverse events from Acalabrutinib with Obinutuzumab | 3 years
  Definitions found in the Common Terminology Criteria for Adverse Events version 5 (CTCAE v 5.0) will be used for grading the severity (intensity) of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Meghan Thompson, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Memorial Sloan Kettering Basking Ridge (All protocol activities), Basking Ridge, New Jersey
  - Hackensack Meridian Health (Data collection only), Hackensack, New Jersey
  - Memorial Sloan Kettering Monmouth (All protocol activities), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (All protocol activities), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (All protocol activities), Commack, New York
  - Memorial Sloan Kettering Westchester (All protocol activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center (All Protocol Activities), New York, New York
  - Memorial Sloan Kettering Nassau (All protocol activities), Uniondale, New York

IPD SHARING:
Plan to Share IPD: Yes
Memorial Sloan Kettering Cancer Center supports the international committee of medical journal editors (ICMJE) and the ethical obligation of responsible sharing of data from clinical trials. The protocol summary, a statistical summary, and informed consent form will be made available on clinicaltrials.gov when required as a condition of Federal awards, other agreements supporting the research and/or as otherwise required. Requests for deidentified individual participant data can be made beginning 12 months after publication and for up to 36 months post publication. Deidentified individual participant data reported in the manuscript will be shared under the terms of a Data Use Agreement and may only be used for approved proposals. Requests may be made to: crdatashare@mskcc.org.

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm